CLINICAL TRIAL: NCT00745758
Title: The Factors Cause Vasospasm After Aneurysmal Subarachnoid Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Kuo-Chuan Wang, Devision of neurosurgery
Other Study IDs: 200803080R
Record Dates: First submitted 2008-08-31; First posted 2008-09-03 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Subarachnoid Hemorrhage; Vasospasm, Intracranial
Keywords: SAH, vasospasm, ADMA
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CSF
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Extensive research has shown that the big event that leads to the initiation of vasospasm is the release of oxyhemoglobin (blood breakdown product).Depletion of NO synthase (19,20,21) was also noted after SAH.CSF is produced from choroid plexus in the ventricle. If the SAH is too dense, the blood in the subarachnoid space will not easy to be washed out.

DETAILED DESCRIPTION:
Cerebral vasospasm remains a significant source of morbidity and mortality in patients with subarachnoid hemorrhage (SAH) after an aneurysmal rupture. Despite being a significant source of morbidity and mortality, death and disability from vasospasm have declined from approximately 35% in the early 1970's, to between 15% and 20% in the 1980's to <10% in the 1990's(1,2,3,4).Extensive research has shown that the big event that leads to the initiation of vasospasm is the release of oxyhemoglobin (blood breakdown product)(1,12,13). This mechanism appears to be a multifactorial process that involves the generation of free radicals, lipid peroxidation and activation of protein kinase C as well as phospholipase C and A2 with resultant accumulation of diacylglycerol and the release of endothelin-1(14,15,16,17,18). On the other hand, depletion of NO synthase (19,20,21) was also noted after SAH. Previous reports showed that shunting of CSF through a lumbar drain after an SAH markedly reduces the risk of clinically evident vasospasm and its sequelae, shortens hospital stay, and improves outcome. Its beneficial effects are probably mediated through the removal of spasmogens that exist in the CSF(22). In our preliminary data, we have demonstrated a case with severe vasospasm, CSF was collected both from EVD and lumbar drain. The ADMA level and amount of Nitrate was well correlate with vasospasm and the level was much higher in lumbar drain then EVD. So, we will compared the CSF from EVD and lumbar puncture to see which factor is correlate with vasospasm.

ELIGIBILITY:
Inclusion Criteria:

* Aneurysmal rupture with SAH

Exclusion Criteria:

* Bleeding tendency,
* Large ICH with impending herniation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient of spontaneous SAH
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-05; Study Completion 2008-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Chuan Wang, MD, Principal Investigator — NTUH
Locations (1):
- devision of neurosurgery, National taiwan university hospital, Taipei, Taiwan